CLINICAL TRIAL: NCT02482532
Title: Phase I Study of Vaccine Enriched, Autologous, Activated T-Cells Redirected to the Tumor Marker GD2 in Patients With Relapsed/Refractory Melanoma
Brief Title: Vaccine Enriched, Autologous, Activated T-Cells Directed to Tumor in Patients With Relapsed/Refractory Melanoma
Acronym: MARVSmALo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gary Doolittle (Other)
Responsible Party: Sponsor-Investigator, Gary Doolittle, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mel-2012-01-01
Record Dates: First submitted 2015-06-18; First posted 2015-06-26 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2021-11

CONDITIONS: Melanoma
Keywords: Melanoma; metastatic; relapsed; refractory
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tvs-CTL Vaccine (Experimental): Infusion of activated T-cells generated from a patient's own peripheral blood mononuclear cells.
  Interventions: Biological: tvs-CTL Vaccine

INTERVENTIONS:
Biological: tvs-CTL Vaccine — autologous, 14g2a.zeta chimeric receptor transduced, activated T-cells, enriched for vaccine specific cytotoxic T-lymphocytes (tvs-CTL)

SUMMARY:
The researchers will investigate if modified T-cells from a patients own system can be utilized to find and destroy metastatic melanoma tumor and thus improve patient outcomes.

DETAILED DESCRIPTION:
The rate of progression free survival at one (1) year is < 20% for patients with stage IV metastatic melanoma, despite aggressive cytotoxic chemotherapy regimens and newly approved immunomodulatory and targeted therapy. Immunotherapy seems to hold the most promise for achieving prolonged survival or even cure, therefore,efforts have focused on several different approaches. Such approaches have used tumor vaccination, adoptive transfer of tumor infiltrating lymphocytes, and even monoclonal antibodies, unconjugated or conjugated to cytokines, toxins, or radionucleotides.

The tumor-associated antigen GD2 has been noted on the surface of several tumors, most notably neuroblastoma, but is expressed on melanoma as well. Clinical studies have shown activity of a GD2-specific chimeric T-cell receptor expressed on activated, autologous, T-cells in patients with neuroblastoma. It is the investigators intention to enrich peripheral blood mononuclear cells (PBMC) of patients with stage IV metastatic melanoma with vaccine-specific T-cells through pre-harvest/ phlebotomy vaccination with common, well understood vaccines. The investigators will then modify the T-cells to attack the GD2 antigen. These tumor redirected, vaccine specific, activated T-cells will then be infused into the patient following revaccination with the common vaccines. The Investigators will monitor expansion of the modified T-cells through serial polymerase chain reaction (PCR) assays following vaccination.

The Investigators then intend to re-vaccinate with the selected vaccines one month following infusion and monitor for expansion of the modified T-cells.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, surgically unresectable melanoma or newly diagnosed melanoma of any stage, where the patient is unable to receive or complete standard therapy
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2
* Laboratory Values

  * absolute neutrophil count > 500 microliters (mcL)
  * platelet > 50,000 mcL
  * serum aspartate aminotransferase (AST) < 5 x institutional upper limit of normal (IULN)
  * total bilirubin < 3 x IULN
  * serum creatinine < 3 x IULN
* Pulse oximetry of > 95% on room air.
* Must have recovered from the toxic effects of all prior chemotherapy

Exclusion Criteria:

* Patients with rapidly progressive disease.
* Patient is currently receiving any investigational drugs
* Current cardiomegaly or bilateral pulmonary infiltrates on chest radiograph, pulmonary metastatic lesions are allowed
* Patients must not have tumor in a location where enlargement could cause airway obstruction
* Patient is pregnant or lactating
* History of hypersensitivity reactions to murine protein-containing products.
* Currently receiving immunosuppressive drugs such as corticosteroids (excluding topical treatment), tacrolimus or cyclosporin
* Received any tumor vaccines within previous six weeks
* Known hypersensitivity to rat monoclonal antibodies
* History of severe allergic reaction to Hepatitis B vaccine, Polio vaccine or Tetanus, Diphtheria, Pertussis vaccine (DTP, Tdap, DT or Td).
* Allergy to baker's yeast or other components of the vaccines.
* History of allergy to the antibiotics Neomycin, Streptomycin or Polymyxin B
* History of coma, long/multiple seizures within 7 days after DTP or Tdap, unless a cause other than the vaccine was indicated.
* Melanoma involvement of the central nervous system
* Chemotherapy given within the last 28 days
* Presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Measurement of infusion related adverse events to evaluate the safety of infused T-cells | 4 weeks
  To evaluate the safety of autologous, receptor-transduced, activated T-cells, enriched for vaccine-specific cytotoxic T-lymphocytes (tvs-CTL)
PCR measurement of retroviral construct to measure persistence of infused T-cells | 4 weeks
  To evaluate how long the infused T-cells remain in the blood stream
Measurement of replication competent retrovirus to evaluate the safety of infused T-cells | 4 weeks
  To evaluate the safety of autologous, receptor-transduced, activated T-cells, enriched for vaccine-specific cytotoxic T-lymphocytes (tvs-CTL)

SECONDARY OUTCOMES:
PCR measurement of retroviral construct to measure the expansion of infused T-cells | 12 months
  To determine the expansion of infused tvs-CTL in response to repeat vaccination with previously administered vaccines
PCR measurement of retroviral construct to compare frequency of peripheral tvs-CTL population pre-infusion vs post-revaccination | 12 months
  To compare the frequency of tvs-CTL in the peripheral blood, after revaccination, to the frequency noted in the prior study of autologous activated, CAR-transduced T-cells infused in patients with relapsed, refractory Stage IV melanoma
Imaging studies to measure tumor response | 10 weeks
  Evaluate tumor response to infusion of tvs-CTL and repeat vaccination post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Doolittle, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- KU Cancer Center, Fairway, Kansas, United States